CLINICAL TRIAL: NCT04401943
Title: Pilot Study of an Online Fatigue Intervention Program for People With Scleroderma
Brief Title: Online Fatigue Intervention Program for People With Scleroderma
Acronym: FAME-ISS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-083
Record Dates: First submitted 2020-05-13; First posted 2020-05-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fatigue intervention (Experimental): the Fatigue intervention is a 6 week intervention delivered using video teleconferencing
  Interventions: Other: online fatigue intervention

INTERVENTIONS:
Other: online fatigue intervention — on line teleconferencing fatigue intervention for 6 weeks on causes of fatigue, ways to protect joint and save energy, ways to manage stress, pain, good eating habits, and exercise.

SUMMARY:
This research is being done to evaluate if an online fatigue intervention program will decrease fatigue, pain and increase confidence managing fatigue and being able to do daily tasks. This study involves competing a series of questionnaires before and after the intervention , and attending and participating in the online videoconference fatigue program for 1 1/2 hour meetings each week over a 6-week period of time.

DETAILED DESCRIPTION:
If eligible and give consent, participants will be asked to complete 2 online questionnaires. The first questionnaire asks basic information such as your age, gender, educational level, and amount of time diagnosed with systemic sclerosis. The second questionnaire asks about your disease symptoms.

You will also be asked to complete questionnaires about your fatigue, pain, mood, confidence in managing your disease and performing daily tasks, and knowledge and use of energy saving techniques.

Once you compete the questionnaires, you will be asked to compete a survey about times and days you would be available to attend the online videoconference fatigue program meeting over a 6 week period of time.

Once the time and dates for the fatigue program are scheduled, you will be expected to attend and take part (using visual and audio) in each 1 ½ hour meeting for 6 weeks online.

The fatigue program includes information on causes of fatigue, ways to protect joint and save energy, ways to manage stress, pain, good eating habits, and exercise. Outside of meetings, you will also be expected to do any "homework" assignments in between the group meetings such as setting goals and doing activities to reach your goals.

At the end of the 6 weeks, you will be asked to complete the same questionnaires you did at the beginning of the study regarding, fatigue, pain, and ability to perform daily tasks. You will also be asked to complete an evaluation of the course.

3 months later, you will be asked to take part in a 45 minute telephone interview to talk about your fatigue and how you are using the ideas from the program.

ELIGIBILITY:
Inclusion Criteria:

* Resident of the United States
* Diagnosis of systemic scleroderma
* 18 years of age or older
* Have use of a device with internet and email access, and video conferencing capabilities (both audio and visual)
* Communicate in English
* Have fatigue (combined score of >12 on 3 questions that rate degree of fatigue, severity of fatigue, and level of stress caused by fatigue on a scale from 1 - 10)
* Be willing and available to complete the study protocol which consists of attending a 1.5 hour virtual meeting once a week for 6 weeks.

Exclusion Criteria:

* Pregnancy
* Not having use of a device with internet, email access, and video conferencing capabilities (both audio and visual)
* Not able to communicate in English
* Score < 12 on the fatigue screening questions
* Not willing or not able to complete the study protocol or participate in the program at the designated times and days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Modified Fatigue Impact Scale at 6 weeks | baseline, 6 weeks
  self report of impact of fatigue on physical, cognitive and psychosocial functioning
Change from baseline Multidimensional Assessment of Fatigue at 6 weeks | baseline, 6 weeks
  Measures four subjective domains of fatigue: degree and severity, amount of distress it causes, timing, and degree to which fatigue interferes with the activities of daily living

OTHER OUTCOMES:
Change from baseline Hospital Anxiety and Depression Scale at 6 weeks | baseline, 6 weeks
  Measures anxiety and depression
Change from baseline PROMIS Self-Efficacy for Managing Symptoms at 6 weeks | baseline, 6 weeks
  Measures participants' confidence in managing symptoms so as not to interfere with the activities they perform in day to day life.
Change from baseline Self-Efficacy for Performing Energy Conservation Strategies Assessment at 6 weeks | baseline, 6 weeks
  Measures participants' confidence in their ability to use energy conservation strategies
Energy Conservations Strategies Survey | 6 weeks
  Measures people's use of energy conservation strategies

CONTACTS AND LOCATIONS:
Overall Officials: Janet L Poole, PhD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carandang K, Poole J, Connolly D. Fatigue and activity management education for individuals with systemic sclerosis: Adaptation and feasibility study of an intervention for a rare disease. Musculoskeletal Care. 2022 Sep;20(3):593-604. doi: 10.1002/msc.1617. Epub 2022 Feb 6. PMID 35124888